CLINICAL TRIAL: NCT00904501
Title: Cell Therapy in Critical Limb Ischemia
Brief Title: Bone Marrow Autograft in Limb Ischemia
Acronym: BALI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHU de Reims (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Principal Investigator, PIGNON, MD, CHU de Reims
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC2007- N11-02
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Peripheral Vascular Diseases
Keywords: Limb ischemia; Cell Therapy
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): A bone marrow harvest (500 mL under general anaesthesia) is performed and BM-MNC are separated and concentrated (30mL). A placebo cell-product (30 mL saline with 4 ml peripheral blood) is implanted and the BM-MNC are cryo-conserved. Only the cell therapy unit, neither the patient, nor the clinician, know whether BM-MNC or placebo is implanted. After 6 months, it is possible to use previously cryo-conserved BM-MNC.
  Interventions: Procedure: Bone marrow harvest
- B (Experimental): A bone marrow harvest (500 mL under general anaesthesia) is performed and BM-MNC are separated and concentrated (30mL) . The BM-MNC are implanted on the same day. Only the cell therapy unit, neither the patient, nor the clinician, know whether BM-MNC or placebo is implanted
  Interventions: Procedure: Bone marrow harvest

INTERVENTIONS:
Procedure: Bone marrow harvest — Implantation of placebo
  Arms: A
Procedure: Bone marrow harvest — Implantation of bone marrow - mononuclear cells
  Arms: B

SUMMARY:
BALI (Bone marrow Autograft in Limb Ischemia) is a randomized double-blind trial comparing implantation of bone marrow - mononuclear cells versus placebo in patients presenting with critical leg ischemia and no surgical option.

The main end point is the survival without major amputation 6 months after implantation.

Biological studies are performed on bone marrow mononuclear cells (BM-MNC) to evaluate their angiogenic properties.

DETAILED DESCRIPTION:
One hundred and ten patients with critical leg ischemia and no surgical option will be included. A bone marrow harvest (500 mL under general anaesthesia) is performed and BM-MNC are separated and concentrated (30 mL) for all included patients. For half of them, the BM-MNC are implanted on the same day whereas the others are implanted with a placebo cell-product (30 mL saline with 4 ml peripheral blood). For these patients the BM-MNC are cryo-conserved. Only the cell therapy unit, neither the patient, nor the clinician, know whether BM-MNC or placebo is implanted. The main end point is the survival without major amputation 6 months after implantation. After this delay it is possible to use previously cryo-conserved BM-MNC. Likewise biological studies are performed on BM-MNC: flow-cytometry analysis of progenitor cells content, proteins and mRNAs expression, induced angiogenesis in animal models.

ELIGIBILITY:
Inclusion Criteria:

* Critical limb ischemia
* No possible surgical treatment

Exclusion Criteria:

* Ongoing infectious disease
* Gangrene extending beyond the digits
* Diabetes mellitus with HbA1c > 7.5% or with proliferative retinopathy
* History of malignant disease
* Contra-indication to general anaesthesia
* Chronic haemodialysis
* Prothrombin Time < 50%
* Recent onset (within 3 months) of myocardial infarction or brain infarction
* Contra-indication to modification of anti-platelet or anticoagulant therapy
* History of heparin-induced thrombocytopenia
* Unexplained haematological abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Major amputation rate and mortality | 6 months

SECONDARY OUTCOMES:
Clinical symptoms and haemodynamical parameters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard PIGNON, Study Director — CHU REIMS FRANCE
Locations (14):
- France (14):
  - CHU, Amiens
  - CHU, Besançon
  - CHU, Bordeaux
  - CHU, Caen
  - CHU, Grenoble
  - CHU, Lille
  - CHU, Limoges
  - CHU, Marseille
  - Centre Hospitalier, Mulhouse
  - CHU, Nancy
  - CHU, Nantes
  - HEGP, Paris
  - Chu Reims, Reims
  - Chu Strasbourg, Strasbourg